CLINICAL TRIAL: NCT00316355
Title: Stepped Care for Obsessive-Compulsive Disorder
Brief Title: Stepped Care for Treating Obsessive-Compulsive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hartford Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, David Tolin, Principal Investigator, Hartford Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R34MH071464 (NIH); R34MH071464 (NIH)
Record Dates: First submitted 2006-04-18; First posted 2006-04-20 (Estimated); Results first posted 2016-06-06 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-01

CONDITIONS: Obsessive-compulsive Disorder
Keywords: Anxiety; Behavior therapy; Cognitive-behavioral therapy; Stepped care; Cost-effectiveness
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Traditional CBT (Active Comparator): Cognitive-behavioral therapy (CBT) that incorporates exposure with ritual prevention (EX/RP)
  Interventions: Behavioral: Traditional CBT
- Stepped-Care CBT (Experimental): Stepped-care CBT
  Interventions: Behavioral: Stepped-Care CBT

INTERVENTIONS:
Behavioral: Traditional CBT — CBT with EX/RP is a psychosocial treatment that incorporates exposure with ritual prevention.
  Arms: Traditional CBT
Behavioral: Stepped-Care CBT — In the CBT stepped-care program, patients are first provided with a less expensive, less intrusive, and more accessible option that resembles quality community care (e.g., self-administered EX/RP combined with counseling to address medication issues, life stress, and motivational enhancement). Patients who fail to respond to this initial treatment progress to a more intensive treatment (e.g., therapist-administered EX/RP).
  Arms: Stepped-Care CBT

SUMMARY:
This study will determine the effectiveness and cost-effectiveness of a stepped-care treatment program for people with obsessive-compulsive disorder.

DETAILED DESCRIPTION:
Obsessive-Compulsive Disorder (OCD) is a chronic and debilitating anxiety disorder. People with OCD often experience recurrent unwanted thoughts, called obsessions, and repetitive behaviors, called compulsions. These thoughts and behaviors interfere with everyday life to a great extent. Currently, the most frequently used psychosocial treatment for OCD is cognitive-behavioral therapy (CBT) that incorporates exposure with ritual prevention (EX/RP). However, although effective, this treatment approach is largely inaccessible, time-consuming, labor-intensive, and expensive. A stepped-care approach to treating OCD may be more cost-effective and therefore more accessible for many individuals. Stepped-care CBT begins with the least expensive, least intrusive, most accessible option, and works up to the most expensive option if the less intrusive treatments do not work. This study will determine the benefits and cost-effectiveness of a stepped care treatment program for OCD.

Participants in this open label study will be randomly assigned to receive CBT for 6 to 14 weeks either through the stepped-care approach or immediately upon study entry. Participants will report to the study site for treatments and assessments on a regular basis, ranging from every 2 weeks to twice a week, depending on the stage of the study and the assigned treatment group. Stepped-care CBT will begin with self-administered EX/RP combined with counseling to address medication issues, life stress, and motivational enhancement. If ineffective, this treatment will be followed by therapist-administered EX/RP. OCD symptoms will be assessed at Week 6. Participants who have responded to treatment after 6 weeks will not receive further treatment. All others will continue for an additional 8 weeks. These participants' OCD symptoms will be assessed again at Week 14. Participants assigned to the stepped-care approach whose OCD symptoms improved initially, but relapsed without further treatment by the Week 14 evaluation will receive full-scale CBT. Outcomes will be assessed again at 1- and 3-month follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of OCD of moderate or greater severity
* Presence of OCD symptoms for at least 1 year

Exclusion Criteria:

* History of psychotic or developmental disorder
* Uncontrolled bipolar disorder
* Serious suicide risk
* Prior history of adequate CBT, including exposure and response prevention

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2006-06; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David F. Tolin, PhD, Principal Investigator — Institute of Living/Hartford Hospital
Locations (1):
- Institute of Living/Hartford Hospital, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tolin, D.F., Diefenbach, G.J., Maltby, N., & Hannan, S. (2005). Stepped care for obsessive-compulsive disorder: A pilot study. Cognitive and Behavioral Practice, 12, 403-414.

RESULTS

PARTICIPANT FLOW:
Groups:
- Traditional CBT: Cognitive-behavioral therapy (CBT) that incorporates exposure with ritual prevention (EX/RP)
  Cognitive-Behavioral Therapy with EX/RP: CBT with EX/RP is a psychosocial treatment that incorporates exposure with ritual prevention.
Period: Overall Study
Arm/Group | Traditional CBT | Stepped-Care CBT
Started | 15 | 19
Started Treatment | 12 | 18
Completed | 10 | 12
Not Completed | 5 | 7

BASELINE CHARACTERISTICS:
Population: Participants randomized to treatment conditions
Groups:
- Total: Total of all reporting groups
Arm/Group | Traditional CBT | Stepped-Care CBT | Total
Number analyzed (Participants) | 15 | 19 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.33 (10.50) | 35.95 (16.16) | 33.74 (13.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 13 | 20
  Male | 8 | 6 | 14
Region of Enrollment [Number; unit: participants]
  United States | 15 | 19 | 34

OUTCOME MEASURES:

1. Primary Outcome: Yale-Brown Obsessive-Compulsive Scale (Y-BOCS) Total Score
Description: The Yale-Brown Obsessive-Compulsive Scale (Y-BOCS) total score was used as the outcome measure. The Y-BOCS is a clinician-rated scale assessing obsession (5 items) and compulsion (5 items) symptom severity on a 0 to 4 scale. All 10 items are added for the total score, with total scores ranging from 0 to 40, and higher numbers indicating more severe symptoms.
Time Frame: Pretreatment, Posttreatment, and 3-month follow-up
Population: Randomized participants
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Traditional CBT | Stepped-Care CBT
Number analyzed (Participants) | 15 | 19
units on a scale
  Pretreatment | 26.00 (5.54) | 24.47 (5.54)
  Posttreatment | 14.25 (6.19) | 15.16 (5.54)
  3-Month Follow-up | 15.75 (6.40) | 13.87 (6.26)

2. Primary Outcome: Treatment-related Total Cost Estimates
Description: total estimated costs calculated based upon the fixed-dose schedule
Time Frame: Posttreatment
Population: Treatment completers
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Traditional CBT | Stepped-Care CBT
Number analyzed (Participants) | 10 | 12
dollars | 5222.80 (1429.15) | 3121.65 (2826.93)

ADVERSE EVENTS:
Arm/Group | Traditional CBT | Stepped-Care CBT
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/18
Other Adverse Events (participants affected / at risk) | 0/12 | 1/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Traditional CBT (N=12) | Stepped-Care CBT (N=18)
increased anxiety impairing functioning (Psychiatric disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No